CLINICAL TRIAL: NCT02442934
Title: A Multicomponent Intervention to Reduce Perceived Discomforts in Critically Ill Patients: a Randomized Controlled Trial
Brief Title: Reducing Discomforts in Critically Ill Patients: the IPREA3 Study
Acronym: IPREA3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Pierre KALFON (Other)
Responsible Party: Sponsor-Investigator, Dr Pierre KALFON, MD, PhD, Centre Hospitalier of Chartres
Organization: Centre Hospitalier of Chartres (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012-AO1696-37
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Critical Illness
Keywords: Critical Care; Critical Care Nursing; Discomfort; Sleep deprivation; Noise; Thirst; Pain
MeSH Terms: conditions — Critical Illness; Sleep Deprivation; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multicomponent program (Experimental): Multicomponent intervention to reduce perceived discomforts in critically ill patients : the IPREA3 program
  Interventions: Other: Administration of the IPREA3 questionnaire; Other: Immediate feedback through electronic reminder messages; Other: Targeted interventions in each ICU to reduce discomforts
- Standard Care (Active Comparator): Standard care
  Interventions: Other: Administration of the IPREA3 questionnaire

INTERVENTIONS:
Other: Administration of the IPREA3 questionnaire — On the day of the ICU discharge, the bedside nurse administers to the patient the 18-item IPREA questionnaire i.e the nurse asks the patient to rate the severity of each discomfort source contained in the IPREA3 questionnaire experienced during the entire stay in the ICU
Other: Immediate feedback through electronic reminder messages — After the nurse had administered the questionnaire, warning messages are displayed on the screen corresponding to the key points to prevent the three discomforts reported with the highest scores
  Arms: Multicomponent program
Other: Targeted interventions in each ICU to reduce discomforts — These targeted interventions are implemented through the coordination of two local champions.
  The central coordination IPREA3 team sends each month to the local champions monthly and cumulative discomfort scores of their unit (overall score of discomfort and scores for each item) and their ranking relative to other units assigned to the interventional arm i.e applying the IPREA3 program.
  The local champions organize monthly meetings with the unit staff to present the results in terms of perceived discomforts measured by the IPREA questionnaire, identify main discomfort sources and actions to be conducted to reduce the discomforts reported with the highest scores in the unit and those that are most easily preventable, and assess the efficacy of already applied measures.
  Arms: Multicomponent program

SUMMARY:
Since critically ill patients are exposed to stressful conditions, the investigators evaluated the effectiveness of a multicomponent program to reduce perceived discomforts in the Intensive Care Unit (ICU) .

DETAILED DESCRIPTION:
The investigators conducted a cluster-randomized trial randomizing 34 ICUs. The program targeted staff members with 3 components : web-based systematic measurement of discomforts on the day of ICU discharge by institutional caregivers (nurses and assistant nurses of the participating ICU), immediate feedback through electronic reminder messages intended to caregivers, and targeted interventions in each ICU based on comparative discomfort scores monthly reported to local champions who were also responsible for staff education.

The measurement of discomforts perceived by critically ill patients at the end of the ICU stay, related to the whole stay in the ICU, was performed by the bedside nurse using a specific questionnaire, the IPREA questionnaire whose construct validity, external validity, reliability, reproducibility and acceptability have been already demonstrated (Development and validation of a questionnaire for quantitative assessment of perceived discomforts in critically ill patients. Kalfon P et al, Intensive care Med 2010, 36:1751-58). The version of the IPREA questionnaire used in the study was a 18-item questionnaire : noise ; excessive light ; discomfort related to sleeping in a different bed from home ; sleep deprivation ; thirst ; hunger ; feeling of cold ; feeling of heat ; pain ; being tied down by perfusion lines, tubes or as a result of connections due to monitoring devices ; no respect for intimacy ; anxiety ; isolation ; limited visiting hours ; absence of phone ; lack of information ; shortness of breath ; and depression.

The duration of the program is 6 months in each arm. Potential participants in the study were consecutive patients admitted in all the participating ICU that are divided in two groups of 17 ICUs.

During October 2014, the IPREA questionnaire is administered to all potentially eligible patients hospitalized in the 34 participating ICUs without applying the program (period P1). The 17 ICUs of the group 1 do not apply the multicomponent program during 5 months (until March 2015), while the 17 ICUs of the group 2 apply the program (period P2). During April 2015, the questionnaire IPREA is administered again in both groups (period P3). From May 2015 until September 2015, the multicomponent program is only applied in the group 1 and no longer in the group 2 (period P4) in order to achieve the crossover of the intervention. During October 2015, the questionnaire IPREA is administered again in both groups (period P5).

The overall score of discomfort and the scores for each item will be compared in the control arm and in the interventional arm.

The control arm consists in the patients included in the group 2 during October 2014 and the patients included in the group 1 during April 2015, i.e. patients included during the month preceding the implementation of the multicomponent program.

The interventional arm consists in the patients included in the group 2 during April 2015 and the patients included in the group 1 during October 2015, i.e. patients included during the last month of the period of application of the multicomponent program.

ELIGIBILITY:
Inclusion Criteria:

* adult critically ill patients
* ICU stay of three calendar days or more

Exclusion Criteria:

* deceased patient in the ICU
* ICU stay of two calendar days or less
* patient younger than 18
* patient under trusteeship
* patient refusing to participate to the study
* patient with diminished mental capacity
* patient not understanding French sufficiently to be questioned (language barrier)
* transfer to another ICU while mechanically ventilated
* emergency discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5411 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Overall score of discomfort | 1 Day of discharge from the ICU
  Each discomfort-item is scored 0-10 (example 0 = no pain ; 10 = pain as bad as can be). For each individual, the overall score of discomfort is computed as the mean of the 18 scores reported for each discomfort-item multiplied by 10, yielding an overall score between 0 and 100.

SECONDARY OUTCOMES:
Scores reported for each discomfort-item | 1 Day of discharge from the ICU
  Each of the 18 discomfort-items is scored 0-10 (example 0 = no thirst ; 10 = thirst as bad as can be).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre KALFON, MD, PhD, Principal Investigator — CH CHARTRES
Locations (26):
- France (26):
  - CH Auxerre, Auxerre
  - Hôpital de la Cavale Blanche, Brest
  - CH Louis Pasteur, Chartres
  - CHU Beaujon APHP, Clichy
  - CHU Hôpital Bocage, Dijon
  - CH Douai, Douai
  - CHU Raymond Poincaré APHP, Garches
  - CH La Rochelle, La Rochelle
  - CH Le Puy en Velay, Le Puy-en-Velay
  - CH Lens, Lens
  - CHU Edouard Herriot, Lyon
  - Hôpital Européen, Marseille
  - CHU Hôpital Nord, Marseille
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - CHU Hôpital Pasteur2, Nice
  - CHU Saint Louis APHP, Paris
  - CHU La Pitié Salpétrière APHP, Paris
  - CHU Cochin APHP, Paris
  - Hôpital Saint Joseph, Paris
  - CHU Hôpital Européen Georges Pompidou APHP, Paris
  - CHU La Milétrie, Poitiers
  - CH Victor Provo, Roubaix
  - CHU NHC, Strasbourg
  - CHU Hautepierre, Strasbourg
  - Hôpital Saint Musse, Toulon
  - CH Troyes, Troyes

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kalfon P, Mimoz O, Auquier P, Loundou A, Gauzit R, Lepape A, Laurens J, Garrigues B, Pottecher T, Malledant Y. Development and validation of a questionnaire for quantitative assessment of perceived discomforts in critically ill patients. Intensive Care Med. 2010 Oct;36(10):1751-1758. doi: 10.1007/s00134-010-1902-9. Epub 2010 May 26. PMID 20502874
- [Derived] Kalfon P, Boucekine M, Estagnasie P, Geantot MA, Berric A, Simon G, Floccard B, Signouret T, Fromentin M, Nyunga M, Audibert J, Ben Salah A, Mauchien B, Sossou A, Venot M, Robert R, Follin A, Renault A, Garrouste-Orgeas M, Collange O, Levrat Q, Villard I, Thevenin D, Pottecher J, Patrigeon RG, Revel N, Vigne C, Azoulay E, Mimoz O, Auquier P, Baumstarck K; IPREA Study Group. Risk factors and events in the adult intensive care unit associated with pain as self-reported at the end of the intensive care unit stay. Crit Care. 2020 Dec 7;24(1):685. doi: 10.1186/s13054-020-03396-2. PMID 33287910
- [Derived] Baumstarck K, Boucekine M, Estagnasie P, Geantot MA, Berric A, Simon G, Floccard B, Signouret T, Fromentin M, Nyunga M, Sossou A, Venot M, Robert R, Follin A, Audibert J, Renault A, Garrouste-Orgeas M, Collange O, Levrat Q, Villard I, Thevenin D, Pottecher J, Patrigeon RG, Revel N, Vigne C, Azoulay E, Mimoz O, Auquier P, Kalfon P; IPREA Study group. Assessment of patients' self-perceived intensive care unit discomforts: Validation of the 18-item version of the IPREA. Health Qual Life Outcomes. 2019 Feb 7;17(1):29. doi: 10.1186/s12955-019-1101-5. PMID 30732654
- [Derived] Kalfon P, Baumstarck K, Estagnasie P, Geantot MA, Berric A, Simon G, Floccard B, Signouret T, Boucekine M, Fromentin M, Nyunga M, Sossou A, Venot M, Robert R, Follin A, Audibert J, Renault A, Garrouste-Orgeas M, Collange O, Levrat Q, Villard I, Thevenin D, Pottecher J, Patrigeon RG, Revel N, Vigne C, Azoulay E, Mimoz O, Auquier P; IPREA Study group. A tailored multicomponent program to reduce discomfort in critically ill patients: a cluster-randomized controlled trial. Intensive Care Med. 2017 Dec;43(12):1829-1840. doi: 10.1007/s00134-017-4991-x. Epub 2017 Nov 27. PMID 29181557
- [Derived] Kalfon P, Mimoz O, Loundou A, Geantot MA, Revel N, Villard I, Amour J, Azoulay E, Garrouste-Orgeas M, Martin C, Sharshar T, Baumstarck K, Auquier P. Reduction of self-perceived discomforts in critically ill patients in French intensive care units: study protocol for a cluster-randomized controlled trial. Trials. 2016 Feb 16;17:87. doi: 10.1186/s13063-016-1211-x. PMID 26880373